CLINICAL TRIAL: NCT00538655
Title: A Pilot Trial of Modafinil for Treatment of Methamphetamine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, Gantt Galloway, PharmD, Scientist, California Pacific Medical Center Research Institute
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 27.004
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Methamphetamine Addiction
Keywords: amphetamine; methamphetamine; addition; treatment study; drug use; modafinil
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- modafinil (Experimental)
  Interventions: Drug: modafinil

INTERVENTIONS:
Drug: modafinil — 400mg vs. 200mg (PO) daily
  Other Names: Provigil

SUMMARY:
Patients treated for methamphetamine dependence have high rates of relapse, and no pharmacotherapy has yet been demonstrated to be efficacious. Modafinil (d, l-2-[(diphenylmethyl) sulfinyl] acetamide) is a novel wake- and vigilance- promoting agent that is chemically and pharmacologically dissimilar to CNS stimulants such as the amphetamines, methylphenidate, and pemoline. It is well tolerated and has low abuse liability compared to CNS stimulants. Modafinil is FDA approved for a variety of sleep disorders, may relieve methamphetamine withdrawal symptoms, improves cognitive function, has been shown to reduce cocaine use in dependent users, and is safe when co-administered with intravenous methamphetamine. We will conduct a pilot, open-label clinical trial of modafinil to establish its safety and efficacy as a pharmacotherapy for methamphetamine dependence.

Specific Aims:

1. Determine the safety of modafinil in the treatment of methamphetamine dependence.
2. Determine the efficacy of modafinil in the treatment of methamphetamine dependence.
3. Assess the effect of modafinil on cognitive function in methamphetamine users.
4. Assess the effect of modafinil on methamphetamine withdrawal symptoms.
5. Compare the validity of a cellular telephone-based reporting system for assessing medication regimen adherence to conventional electronic medication monitoring.

Hypotheses:

1. Modafinil will be as safe and well tolerated as placebo in a comparison group from another study.
2. Subjects given modafinil will use less methamphetamine than subjects given placebo.
3. Subjects given modafinil with demonstrate improvements in cognitive function when compared to subjects given placebo.
4. Subjects given modafinil will have reduced withdrawal symptoms when compared to subjects given placebo.
5. Adherence will be recorded more accurately by cellular telephone than by conventional electronic medication monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Patient is agreeable to conditions of study and signs consent form
* Fluency in English

Contact site for additional information.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
MA (-) urine samples | multiple

CONTACTS AND LOCATIONS:
Overall Officials: Gantt Galloway, Pharm D., Principal Investigator — California Pacific Medical Center
Locations (1):
- CPMC - St. Luke's Hospital ~ 7th Floor/ Addiction Pharmacology Research Lab, San Francisco, California, United States